CLINICAL TRIAL: NCT05998252
Title: A Post-Market Study to Evaluate Safety and Efficacy of Alveo HP Balloon Dilatation Catheter for Balloon Dilatation of Coronary Artery Stenosis
Brief Title: Evaluate Safety and Efficacy of Alveo HP Balloon Dilatation Catheter for Balloon Dilatation of Coronary Artery Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BrosMed Medical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S01
Record Dates: First submitted 2023-02-12; First posted 2023-08-18 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alveo balloon dilatation catheter (Experimental): Subjects who meet the inclusion criteria and agree to participate in the study will be enrolled and undergo a planned percutaneous coronary intervention with Alveo balloon dilatation catheter.
  Interventions: Device: Alveo HP Balloon Dilatation Catheter

INTERVENTIONS:
Device: Alveo HP Balloon Dilatation Catheter — Alveo HP Balloon is intended for dilatation of stenosis in the coronary artery.

SUMMARY:
This is a prospective, multi-center, single-group study aims to evaluate the safety and efficacy of Alveo HP Balloon Dilatation Catheter for balloon dilatation of coronary artery stenosis. Pre-dilation with Alveo balloon dilatation catheter followed by conventional PCI, and follow-up will be carried out. During the trial, the enrollment, treatment and follow-up of the subjects will be recorded, and the safety and efficacy of the investigational device will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, gender is not limited;
2. Patients with symptomatic ischemic heart disease who are suitable for percutaneous coronary intervention (PCI);
3. Patients with target lesion diameter stenosis ≥ 70% (visually) or chronic total occlusion (CTO) who needed balloon dilatation catheter pre-dilatation;
4. Patients or their guardians who can understand the purpose of the trial, voluntarily participate and sign the written informed consent, and can accept follow-up;

Exclusion Criteria:

1. Patients with clinical symptoms consistent with ST-segment elevation myocardial infarction or/and ECG changes within 12 hours prior to the procedure;
2. Patients who are known to be intolerant to antiplatelet drugs or allergic to contrast media;
3. Patients with in-stent restenosis;
4. Patients with unprotected left main coronary artery disease;
5. Patients who plan to treat 3 or more lesions at the same time;
6. Patients with severe calcified lesions;
7. Patients in whom the guidewire cannot pass through the lesion;
8. Women who are pregnant or lactating;
9. Patients who are participating in the clinical trial of other drugs or medical devices;
10. Other patients considered by the investigator to be unsuitable for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Procedural Success Rate | 7 days
  Defined as meeting all the following criteria:
  1. After PCI, the target lesion achieves a final diameter stenosis of ≤30%, and the TIMI grade of 3;
  2. No all-cause mortality, Q-wave myocardial infarction, stroke, cardiac tamponade, or target vessel revascularization (including re-PCI or emergency coronary artery bypass grafting) during postoperative follow-up.

SECONDARY OUTCOMES:
Device Success Rate | 0 day
  Defined as meeting all the following criteria:
  1. Successful delivery to the target location, completely pre-dilatation and successful withdrawal by using Alveo HP Balloon Dilatation Catheter;
  2. No evidence of arterial perforation, flow-restricted dissection, decreased TIMI grade while using the device, or no clinically significant arrhythmias after pre-dilatation.
Device Performance Evaluation | 0 day
  The investigators will evaluate the device performance according to the use and operation of the device during the procedure. Evaluate performance of balloon catheter delivery, inflation, deflation, and withdrawal, etc. There are 5 levels ranging from poor to excellent, higher scores indicate better performance.

OTHER OUTCOMES:
Incidence of major adverse cardiac events (MACE) during the study. | 0 - 7 days
  Major adverse cardiac events (MACE) are defined as cardiac death, myocardial infarction, and target lesion revascularization (TLR).
Adverse events and serious adverse events rate | 0 - 7 days
  Adverse events and serious adverse events related to the study device during the study.
Other Adverse events and serious adverse events rate | 0 - 7 days
  Occurrence of other adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Seventh People's Hospital of Zhengzhou, Zhenzhou, Henan
  - Renmin Hospital of Wuhan University Hubei General Hospital, Wuhan, Hubei
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No